CLINICAL TRIAL: NCT04645225
Title: Clinical Characteristic and MEFV Gene Mutations in Patient With Juvenile Onset- Systemic Lupus Erythematosus
Brief Title: Clinical Characteristic and MEFV Gene Mutations in Patient With Juvenile Onest Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shrouk Ahmed Mostsfa Sayed, Resident pediatric, Assiut University
Other Study IDs: MEFV gene in jSLE
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: SLE (Systemic Lupus)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: . MEFV genetic testing — For mutation analysis, 2 ml blood will be with drawn from both patient and control groups in order to obtain genomic DNA. Extraction of DNA molecule from peripheral blood lymphocytes will be done using standard procedures, then amplification of MEFV gene will be done by polymerase chain reaction(PCR). Reversed hybridization technique will be used for identification of MEFV gene mutation.

SUMMARY:
Aim and objectives of this study

* To summarize the main clinical characteristics of patients with jSLE admitted and followed up in Assiut University children's Hospital.
* To compare the MEFV gene mutations in patients with jSLE versus a control group of healthy children in upper-Egypt a country with a considerably high carrier rate for the MEFV gene variants.
* To assess the prevalence and clinical significance of jSLE patients carrying MEFV variants and assess the impact of MEFV gene mutation on disease severity as assessed by systemic lupus erythematous disease activity index (SLEDAI).
* To assess if there is a specific MEFV gene mutations that are more associated with jSLE and/or certain disease manifestations, such as serositis

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune inflammatory disease characterized by the presence of multiple auto antibodies and is associated with a multisystemic illness. The clinical presentation of SLE ranges from mild to severe and the course of the disease is unpredictable, with periods of remission and flares. (1) Juvenile-onset systemic lupus erythematosus (jSLE) patients present more frequently in teenage years and accounts for 15%-20% of lupus population, and they typically have severe disease course than adult patients. A considerable number of jSLE patients have significant renal or central nervous system(CNS) involvement at the time of diagnosis.(1) It is slightly more common in girls, with a sex ratio about 4:3 before puberty; however after puberty, the sex difference increases to about 4:1.(2) The disease is more common in Native Americans,African Americans, and Asians. (3) Prevalence rate of jSLE have varied from 4-250 per 100,000 population.(4,5) JSLE is not rare in Egypt and Africa, representing an important subset that is commonly overlooked and requires special attention. (6,7) SLE ranges from an insidious, slowly progressive, chronic disease with exacerbations and remissions,to an acute and rapidly fatal disease. Constitutiona lfeatures such as fever, fatigue, anorexia, myalgia,weight loss are common both at onset and during exacerbations of the disease. (8,9) Familial Mediterranean fever (FMF), an autosomal recessively inherited autoinflammatory disorder, is characterized by recurrent, self-limited inflammatory attacks involving mainly serosal membranes. The disease has been associated with variations in the MEFV gene, which encodes the pyrin protein, in the great majority of patients.(10) FMF is the most common autoinflammatory disorder, and the rate of heterozygous carrier for MEFV gene variations is quite high in Eastern Mediterranean countries, including Turkey, Israel, and Armenia.(11,12) A higher acute phase response has been reported in asymptomatic heterozygous carriers, and heterozygosity for MEFV variations has been suggested to affect the course of other autoinflammatory disorders.(13,14) A connection between FMF and collagen diseases were suggested previously by multiple studies as that MEFV mutations M694V and M680I were observed to be associated with Behcet's Disease (BD), (15)Also the MEFV variants in exon 10 were suggested to affect the clinical presentation of Henoch-Schönleinpurpurain populations where FMF is common. (16) The mutation p.M694V/I in MEFV gene might be a risk factor for systemic onset juvenile idiopathic arthritis sJIA, (17)and M694V is accepted to be associated with more severe inflammation as compared to other mutations in patients with Polyarteritis nodosa.

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrollment ≤18 years old but they should be diagnosed as jSLE before the age of 16 years old.
2. Both sexes
3. The Patients should be diagnosed as jSLE according to 2019 European league against rheumatism (EULAR)/ American college of rheumatology (ACR) SLE classiﬁcation criteria, (20) or previous ACR 1997 SLE classification criteria.
4. No suggestive symptoms of FMF as stated by Tel Hashomer criteria

Exclusion Criteria:

* 1- Patients diagnosed as FMF or receiving colchicine for possibility of FMF. 2- Patients with other autoimmune disease. 3- Patients not fulfilling the criteria for diagnosis of SLE

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sixty patients diagnosed and followed up as jSLE will be consecutively recruited from the inpatient and outpatient clinic of Immunology and rheumatology department at Assuit University children's hospital. A control group of 40 age and sex matched control will be recruited from the surgery outpatient clinic or relatives of the patients. The study will be conducted during from Jan 2021 to Jan 2022.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
MEFV gene mutations in jSLE | baseline
  compare the MEFV gene mutations in patients with jSLE versus a control group of healthy childrenin upper-Egypt a country with a considerably high carrier rate for the MEFV gene variants

REFERENCES:
- [Background] Tucker LB, Uribe AG, Fernandez M, Vila LM, McGwin G, Apte M, Fessler BJ, Bastian HM, Reveille JD, Alarcon GS. Adolescent onset of lupus results in more aggressive disease and worse outcomes: results of a nested matched case-control study within LUMINA, a multiethnic US cohort (LUMINA LVII). Lupus. 2008 Apr;17(4):314-22. doi: 10.1177/0961203307087875. PMID 18413413
- [Background] Serdula MK, Rhoads GG. Frequency of systemic lupus erythematosus in different ethnic groups in Hawaii. Arthritis Rheum. 1979 Apr;22(4):328-33. doi: 10.1002/art.1780220403. PMID 426879